CLINICAL TRIAL: NCT00847249
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled AZD9164 After Single Ascending Doses in Healthy Male Subjects
Brief Title: AZD9164 Single Ascending Dose Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Anders Luts, Medical Science Director, Emerging Project, Team 3, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1882C00001; EudraCT No.2008-007188-18
Record Dates: First submitted 2009-02-12; First posted 2009-02-19 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: safety; tolerability; healthy; inhalation; Healthy males
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD9164

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Solution for nebulisation, inhaled
  Interventions: Drug: AZD9164
- 2 (Placebo Comparator): Solution for nebulisation, inhaled
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9164 — Each subject will receive a single-dose starting dose 4µg (lung deposited dose) with up to 8 dose escalations not exceeding AstraZeneca pre-defined exposure limits.
  Arms: 1
Drug: Placebo — Each subject will receive a single-dose.
  Arms: 2

SUMMARY:
The aims of the study are to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of AZD9164 following single ascending dose administrations to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically significant abnormalities at screening examinations
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2009-02; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | up to 48 hours post-dose.

SECONDARY OUTCOMES:
Pharmacokinetics | up to 48 hours post-dose.
Local and extrapulmonary effects | up to 48 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Luts, Study Director — AstraZeneca; Ulf Malmqvist, Principal Investigator — Clinical Trial Unit, Clinical Research and Trial Centre, Lund University Hospital, Lund, Sweden
Locations (1):
- Research Site, Lund, Sweden